CLINICAL TRIAL: NCT03702829
Title: 24 Month Open Label Study of the Tolerability and Efficacy of an Antisense Oligonucleotide (Inotersen) in Patients With Transthyretin (TTR) Amyloid Cardiomyopathy
Brief Title: 24 Month Open Label Study of the Tolerability and Efficacy of Inotersen in TTR Amyloid Cardiomyopathy Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Rodney H. Falk, MD, Director, Brigham and Women's Cardiac Amyloidosis Program, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P001436
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Amyloidosis
Keywords: wild-type transthyretin amyloidosis; TTR amyloidosis; familial amyloid cardiomyopathy; mutant transthyretin amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Inotersen; Oligonucleotides, Antisense

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Drug (Experimental): Inotersen, a transthyretin (TTR) antisense oligonucleotide. Administered subcutaneously weekly. Each dose shall contain 300 mg of active drug. Subsequent visits will occur at 3, 6, 12, 18 and 24 months. Every 2 weeks, blood will be monitored for renal function and platelet count and urine will be tested by dipstick for proteinuria.
  Interventions: Drug: Inotersen

INTERVENTIONS:
Drug: Inotersen — Open Label Study
  Other Names: Antisense Oligonucleotide

SUMMARY:
Transthyretin is a protein produced in the liver that transports thyroid hormone and vitamin A. A single substitution of an amino acid in the structure of TTR can result in a relatively unstable protein, the breakdown products of which (predominantly monomers) aggregate abnormally and produce proteinaceous deposits in nerves and the heart. These deposits are known as amyloid and produce progressive nerve and heart damage. Amyloidosis due to a mutant TTR is usually an autosomal dominant and hence is a familial condition. Wild-type TTR is also capable of producing amyloid deposits which predominantly involves the heart (rather than the nervous system) resulting in a progressive decrease in cardiac function with increasing signs of heart failure. This study aims to determine whether subcutaneous injection of an antisense oligonucleotide drug, known as inotersen, that has been specifically designed to reduce production of the protein transthyretin by the liver, can slow or stop the progression of TTR amyloid cardiomyopathy as compared to historical controls, using advanced echocardiography and cardiac MRI. The study also aims to determine the tolerability and safety of this drug when administered over a 24-month period to patients with TTR amyloid cardiomyopathy.

DETAILED DESCRIPTION:
This is an open-label, single center study of 50 patients with cardiac amyloidosis due to wild-type or mutant TTR. Eligible patients will have evidence of cardiac amyloidosis due to transthyretin. The diagnosis will be made by biopsy of the heart or other affected organ with appropriate staining techniques confirming that the amyloid deposits are derived from transthyretin. Alternatively, recent imaging data have shown that a strongly positive nuclear scan using technetium pyrophosphate in the absence of evidence of a plasma cell dyscrasia and in the presence of a typical echocardiographic or cardiac magnetic resonance appearance of cardiac amyloidosis is indicative of TTR amyloidosis and that a biopsy is not needed. This will be acceptable for study entry. As inotersen has been associated with kidney toxicity in a small number of patients, all subjects in the study will be required to have a glomerular filtration rate greater than 45. Once study criteria have been met, and baseline imaging including echocardiography and (where feasible) cardiac magnetic resonance imaging have been performed, all patients will receive inotersen in a weekly 300 mg dosing. Subsequent visits will occur at 6 weeks, and 3, 6, 12, 18 and 24 months. Every 2 weeks, blood will be monitored for renal function and platelet count and urine will be tested by dipstick for proteinuria. Should kidney function be noted to be deteriorating or should proteinuria be found, a more intense renal workup will be performed in order to detect or rule out potential kidney toxicity. At each visit, in addition to standard laboratory work and pregnancy testing if applicable, (complete blood count, comprehensive metabolic panel, thyroid function tests, and urinalysis), Vitamin A level will be drawn (as TTR is a transport protein for Vitamin A) and TTR (prealbumin) level will be drawn to determine degree of suppression. Disease progression will be measured by serial cardiac biomarkers, 6-minute walk, cardiopulmonary stress testing, advanced "strain" echocardiography and cardiac MRI. Patients will be compared to data derived from a historical control group and from data in the literature to determine whether inotersen slows or stops disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have ATTR amyloidosis, defined as is defined as an echocardiographic appearance of left ventricular wall thickness of 13 mm or more, in the absence of uncontrolled hypertension, and with EITHER a positive biopsy for amyloid, which also stains positive for TTR by immunochemistry or mass spectrometry OR a positive cardiac technetium pyrophosphate scan with isotope uptake in the heart equal or greater to rib uptake and with no evidence of a plasma cell dyscrasia.
* For patients meeting the above criteria, wild-type TTR amyloidosis (ATTRwt)will be defined as having transthyretin genetic sequencing negative for a mutation. Mutant/hereditary TTR (ATTRh) will be defined as TTR amyloid cardiomyopathy with TTR sequencing showing an amyloidogenic mutation. A positive biopsy can be from any organ, providing that the echocardiographic appearance is typical of amyloidosis.
* Patients should, in the opinion of the Investigator, be in a stable state in terms of NYHA class. Class I-III patients will be recruited.
* Age 18-85 years
* Male, or non-pregnant, non-lactating females. If a woman is premenopausal, or male partners with a premenopausal woman, she/he must be willing to use the following methods of contraception: condoms, oral/hormonal contraception, intrauterine device, diaphragm, or abstinence
* Written informed consent to be obtained prior to study treatment
* If diagnosis is made by tissue biopsy histochemical diagnosis (positive stains for TTR in absence of staining for light chains, or AA amyloid) in the presence of green birefringent material in Congo red-stained tissue specimens or sulfated Alcian blue stain typical for amyloid deposition. NB. All patients will have had a definitive diagnosis of TTR amyloidosis made prior to study entry, either by tissue biopsy or positive PYP scan, and all will have been genotyped. No further diagnostic testing will need to be done at or after study entry.
* If diagnosis is made by nuclear imaging, a positive technetium pyrophosphate scan, characterized by isotope uptake in the heart of an intensity equal to or greater than, rib uptake.
* Willingness to return to the treating center for follow-up.
* Willingness and ability to self-administer, or to have spouse administer weekly subcutaneous injections of study drug.
* Willingness to take daily oral Vitamin A supplementation throughout the study and for 3 months thereafter.

Exclusion Criteria:

* Patients who, in the opinion of the Investigator, require further adjustment of diuretics at the time of screening to achieve optimal treatment of heart failure. Once stable for 2 weeks, patients in Class I-III will become eligible for inclusion.
* Patients with NYHA class 4 congestive heart failure despite optimal heart failure management.
* Concomitant non-amyloid heart disease that might, in the opinion of the investigator, cause changes in strain imaging on serial follow-up (e.g. aortic stenosis of greater than mild severity, unstable coronary artery disease), or ongoing non-cardiac disease that, in the opinion of the investigator, will likely need hospitalization over the next 2 years (e.g. active cancer) .
* Prior liver transplantation or liver transplantation anticipated in less than 6 months
* ALT and/or AST 2 x ULN and/or Alkaline phosphatase 2 x UNL; Or bilirubin greater than 1.5 times UL (patients with bilirubin ≥1.5 x ULN may be allowed on study if indirect bilirubin only is elevated, ALT/AST is not greater than the ULN and genetic testing confirming Gilbert's disease)
* Glomerular filtration rate (EGFR) < 45 ml/min/1.73m2
* A history of glomerulonephritis,
* Proteinuria or hematuria as detailed in the section below (immediately following exclusion criteria) entitled "Additional information regarding renal exclusion criteria".
* Platelets less than 125×109/L
* TSH values outside normal range in subjects untreated for thyroid disease, unless mildly elevated with normal T4, and deemed by current standards not to need treatment.
* Uncontrolled hypertension (blood pressure >160/100)
* Acute coronary syndrome or major surgery within 3 months of screening
* Anticipated survival less than 2 years
* Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to first dose of study drug
* Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or prostate that has been successfully treated
* Positive test result for HIV, hepatitis B, or hepatitis C
* Any other lab values that in the opinion of the investigator might place the subject at unacceptable risk for participation in the study
* History of poor compliance with medications or medical treatment, based on a review of medical records.
* History of hypersensitivity to any of the ingredients of the study therapy
* Use of any investigational drug for amyloidosis within 4 weeks prior to study entry or during the study.
* Current use of tafamidis, diflunisal, doxycycline or TUDCA for therapy of amyloidosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Systolic strain imaging by echocardiographic | Month 6
  The primary echocardiographic parameter to be measured will be longitudinal left ventricular (LV) strain (units = % LV longitudinal shortening) as compared to baseline.

SECONDARY OUTCOMES:
Systolic strain evaluation by echocardiography | Month 12
  The primary echocardiographic parameter measured will be longitudinal left ventricular (LV) strain (units = %).
Systolic strain evaluation by echocardiography | Month 18
  The primary echocardiographic parameter measured will be longitudinal left ventricular (LV) strain (units = %).
Systolic strain evaluation by echocardiography | Month 24
  The primary echocardiographic parameter measured will be longitudinal left ventricular (LV) strain (units = %).
LV mass measurement by Cardiac MRI (cMRI) (units = grams) | Month 6
  measurement of LV mass by CMR mapping techniques
LV mass measurement by Cardiac MRI (cMRI) (units = grams) | Month 12
  measurement of LV mass by CMR mapping techniques
LV mass measurement by Cardiac MRI (cMRI) (units = grams) | Month 24
  measurement of LV mass by CMR mapping techniques
ECV-extracellular volume by Cardiac MRI (cMRI) (unit=percentage) | Month 6
  measurement of extracellular volume by CMR T1 mapping techniques
ECV-extracellular volume by Cardiac MRI (cMRI) (unit=percentage) | Month 12
  measurement of extracellular volume by CMR T1 mapping techniques
ECV-extracellular volume by Cardiac MRI (cMRI) (unit=percentage) | Month 24
  measurement of extracellular volume by CMR T1 mapping techniques

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Falk, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No